CLINICAL TRIAL: NCT01877681
Title: Chronic Wounds Reference Nurse and Telematic Interconsultation Program for Pressure Ulcers in Primary Care: Evaluation of Effectiveness and Cost Reduction
Brief Title: Reference Nurse Program for Pressure Ulcers in Primary Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Cristina Quesada, Nurse, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011111099
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assisted Care (Experimental): Assisted care (Tele=assistance) provided by an expert nurse through a informatic online application
  Interventions: Procedure: Tele-assistance
- Active comparator (Active Comparator): Usual care as stated by the Clinical Practice Guidelines for Pressure Ulcers treatment
  Interventions: Procedure: Active comparator

INTERVENTIONS:
Procedure: Tele-assistance — Assisted care (Tele-assistance) provided by an expert nurse through a informatic online application
  Arms: Assisted Care
Procedure: Active comparator — Usual care as specified in the PU practice guideline
  Arms: Active comparator

SUMMARY:
Introduction: Pressure ulcers (PU) are the most common chronic wounds in all levels of care in health centers. The chronic wound care by skilled personnel is key to healing and management of these injuries. An inter-clinical telematic program for PU in Primary Care (PC) can improve the effectiveness of interventions and cost savings.

Objective: To evaluate the effectiveness and costs reduction after the implementation in PC setting of a chronic wounds reference nurse and a teleconsultation program aimed to nurses for the management of PU in patients in home care setting.

Methodology: A prospective pilot clinical trial in which 46 primary care nurses in Osakidetza will be randomly assigned to two parallel groups: experimental group and control group. Each nurse will recruit at least 1 new patient in home care with PU in stage II-III. The intervention will consist of a telematic advice from the reference nurse regarding chronic wound management in relation to a specific PU. Patients will be monitored for 8 weeks with a minimum of 4 repeated measurements of the Resvech Index 2.0. To evaluate the effectiveness of the intervention, multilevel models or linear mixed models to take into account the auto-correlation at the individual level and nurse, will be used

ELIGIBILITY:
Inclusion Criteria:

* New cases of PU in Stage II-III, treated by the same nurse over time at patient's home. (Stage II: Partial loss of skin thickness that affects the epidermis, dermis, or both. Ulcer surface that looks like abrasion, blister, or shallow crater; Stage III: Full thickness loss of skin involving damage or necrosis of subcutaneous tissue that may extend down to but not through the underlying fascia)

Exclusion Criteria:

* Patients with chronic wounds that are not PU
* PU in patients with plastic surgery
* Patients who move periodically
* Patients requiring hospitalization during follow-up
* Patients in which nurse is expected to be changed during follow-up
* Terminal patients

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
healing progression | 8 weeks
  healing progression as measured by the RESVECH scale by a blinded expert

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Quesada, Nurse, Principal Investigator — Osakidetza